CLINICAL TRIAL: NCT03596879
Title: Insomnia and Rumination in Late-pregnancy and the Risk for Postpartum Depression (PPD): A Randomized Controlled Trial of Online Cognitive Behavioral Therapy for Insomnia to Prevent PPD
Brief Title: Insomnia and Rumination in Late Pregnancy and the Risk for Postpartum Depression
Acronym: PPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, David Kalmbach, Bioscientific Staff Researcher, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12204
Record Dates: First submitted 2018-06-08; First posted 2018-07-24 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: Insomnia; Post Partum Depression
Keywords: insomnia; post partum depression (PPD); digital CBTI (dCBTI); online CBTI; rumination
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression, Postpartum; Rumination Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dCBTI (Experimental): Online access to the digital CBTI program Sleepio.
  Interventions: Behavioral: dCBTI
- Sleep Education (Placebo Comparator): Weekly email messages with sleep hygiene recommendations.
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: dCBTI — Online access to the digital CBTI program Sleepio based off of traditional face-to-face Cognitive Behavioral Therapy, six weekly sessions done online.
  Arms: dCBTI
Behavioral: Sleep Education — Six weekly email messages with sleep hygiene recommendations. Subjects are encouraged to read through the information and apply it to their sleep.
  Arms: Sleep Education

SUMMARY:
The primary objective of the proposed research is to determine whether prenatal insomnia and ruminative thinking predict severity of postpartum depression (PPD) symptoms. Additionally, the investigators will also determine the effectiveness of digital/internet-based Cognitive Behavioral Therapy for Insomnia (dCBTI) in reducing the risk for PPD.

DETAILED DESCRIPTION:
The purpose of this study is to 1) explore the relationship between prenatal insomnia, ruminative thinking and the severity of PPD symptoms. and 2) determine the effectiveness of Digital Cognitive Behavioral Therapy (dCBTI) in reducing the risk for postpartum depression in pregnant mothers entering into their third trimester. dCBTI is an online form of Cognitive Behavioral Therapy (CBT) that is used with people who experience trouble sleeping at night (insomniacs). As pregnant women are especially vulnerable to sleep problems during this period, this study will help us determine whether dCBTI is helpful in improving sleep and reducing the risk for PPD in this population.

Pregnant women entering their third trimester will be recruited from the Henry Ford Health System through the HFHS Electronic Medical Record (EPIC). They will receive an email from study personnel describing the study, and encouraged to schedule a phone call to discuss study details. Participants will then complete a consent and an online screening survey. Upon meeting inclusion criteria, participants will complete weekly surveys and randomized into one of 2 active online insomnia treatment conditions. Each treatment involves 6 weekly "sessions" which each take up to 20 minutes to complete.

Subjects will complete weekly online surveys beginning at week 30 of pregnancy, and continuing through 6 weeks after giving birth.

ELIGIBILITY:
Inclusion Criteria:

* Must be entering their 3rd trimester of pregnancy
* Must deny any concerns or indications of a high risk pregnancy associated with increased risk for the mother or fetus for negative health outcomes

Exclusion Criteria:

* Age < 18 years old
* Bipolar or seizure disorders (due to risk in CBTI)
* Known sleep disorders other than insomnia (eg narcolepsy, restless legs syndrome, obstructive sleep apnea)
* Women already in their 3rd trimester
* Women who are not pregnant
* Women with high risk pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Improvement in Sleep - Insomnia Severity Index | Year 1
  The Insomnia Severity Index (ISI) is a commonly used self-report measure of insomnia symptoms that has been validated for use in community samples and clinical trials. The ISI scores range from 0-28, with a higher score indicating a greater severity of insomnia.
Prevention of Postpartum Depression Symptoms - Edinburg Postnatal Depression Scale (EPDS) | Year 1
  The Edinburgh Postnatal Depression (EPDS) is the most widely used depression measure in both pregnant and postnatal women. It is validated for use in community samples and clinical trials. The EPDS scores range from 0-30, with a higher score indicating a greater severity of depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Medical Center, Novi, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kalmbach DA, Cheng P, Roth T, Swanson LM, Cuamatzi-Castelan A, Roth A, Drake CL. Examining Patient Feedback and the Role of Cognitive Arousal in Treatment Non-response to Digital Cognitive-behavioral Therapy for Insomnia during Pregnancy. Behav Sleep Med. 2022 Mar-Apr;20(2):143-163. doi: 10.1080/15402002.2021.1895793. Epub 2021 Mar 15. PMID 33719795
- [Derived] Kalmbach DA, Cheng P, O'Brien LM, Swanson LM, Sangha R, Sen S, Guille C, Cuamatzi-Castelan A, Henry AL, Roth T, Drake CL. A randomized controlled trial of digital cognitive behavioral therapy for insomnia in pregnant women. Sleep Med. 2020 Aug;72:82-92. doi: 10.1016/j.sleep.2020.03.016. Epub 2020 Mar 21. PMID 32559716
- [Derived] Kalmbach DA, Cheng P, Ong JC, Ciesla JA, Kingsberg SA, Sangha R, Swanson LM, O'Brien LM, Roth T, Drake CL. Depression and suicidal ideation in pregnancy: exploring relationships with insomnia, short sleep, and nocturnal rumination. Sleep Med. 2020 Jan;65:62-73. doi: 10.1016/j.sleep.2019.07.010. Epub 2019 Jul 22. PMID 31710876